CLINICAL TRIAL: NCT00955916
Title: A Phase II Study of CLAG Regimen in Combination With Imatinib Mesylate (Gleevec) in Relapsed or Refractory Acute Myeloid Leukemia
Brief Title: CLAG Gleevec in Relapsed or Refractory Acute Myeloid Leukemia (AML)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-15787; CSTI571AUS235 (Other: Novartis)
Record Dates: First submitted 2009-08-05; First posted 2009-08-10 (Estimated); Results first posted 2014-01-14 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-06

CONDITIONS: Leukemia
Keywords: relapsed; refractory; acute; myeloid; AML; CML; blast crisis
MeSH Terms: conditions — Leukemia; Recurrence; Blast Crisis | interventions — Cladribine; Cytarabine; Filgrastim; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CLAG Regimen with Gleevec® (Experimental): Combined chemotherapy treatment (CLAG regimen) with Gleevec® (imatinib mesylate).
  Interventions: Drug: CLAG Regimen; Drug: Gleevec®

INTERVENTIONS:
Drug: CLAG Regimen — The CLAG regimen consisted of: Cladribine, 5 mg/m^2 administered via 2 hour IV daily for 5 consecutive days starting on day 2; Cytarabine, 2 mg/m^2 administered through a 4 hour IV starting 2 hours after the ignition of Cladribine for 5 days starting on day 2; granulocyte colony-stimulating factor (G-CSF): 300 mcg subcutaneous (SC) for 6 days starting 12-24 hours (Day 1) before the first dose of Cladribine.
  Other Names: cladribine; cytarabine; neupogen
Drug: Gleevec® — Imatinib mesylate 400 mg orally twice daily was administered on day 2 to day 15. Re-induction was allowed if participant had partial response (PR).
  Other Names: imatinib mesylate

SUMMARY:
The purpose of the study is to find out what effects (good and bad) Gleevec® (Imatinib mesylate) combined with chemotherapy has on participants and their acute myeloid leukemia.

DETAILED DESCRIPTION:
In relapsed or resistant acute myeloid leukemia (a type of blood cancer where immature blood cells are increased, blocking normal blood cell production), different types of chemotherapy are used for treatment. Patients responded to all the chemotherapies in similar ways, but most of the responses did not last long if further stem cell transplantation was not done. Gleevec is believed to work by interfering with the abnormal protein by blocking it from telling the body to keep making more white blood cells that are abnormal.

The CLAG regimen is the standard chemotherapy used for relapsed AML (Acute Myeloid Leukemia). This study will add Gleevec® to the regimen for a period of 14 days. Gleevec® is approved by the Food and Drug Administration (FDA) for the treatment of chronic myeloid leukemia (CML) and some types of acute lymphoblastic leukemia (ALL). Its use in combination with CLAG regimen is considered experimental for the treatment of Acute Myeloid Leukemia/CML blast crisis.

ELIGIBILITY:
Inclusion Criteria:

* Men and Women of all ethnic groups whose age is ≥ 18 years old.
* Diagnosis of AML or CML blast crisis, according to World Health Organization (WHO) criteria, except acute promyelocytic leukemia AML-M3 French-American-British (FAB) subgroup. A documentation of relapse is required by a bone marrow/aspirate within 4 weeks of registration.
* Refractory or Relapsed AML. Refractory AML is defined as failure to achieve CR after 2 cycles of induction chemotherapy or persistent (>40%) bone marrow blasts after one cycle of chemotherapy induction.
* Relapsed AML is defined as any evidence of disease recurrence after achieving complete response (CR) (more than 5% myeloblasts). Early relapse is defined as that occurring within 12 months and late relapse is defines as that occurring after 12 months.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Patients must sign a written informed consent.
* Females of childbearing potential (FOCP) must not be pregnant or actively nursing a child. They must have a negative pregnancy test 7 days before initiation of study drug administration
* Postmenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential.
* Male and females of reproductive potential must agree to employ an effective barrier method of birth control throughout the duration of the trial and for 3 months following study medication discontinuation.
* Prior allogeneic or autologous stem cell transplantation is allowed.

Exclusion Criteria:

* Abnormal Kidney Functions: creatinine ≥2.5 mg/dL.
* Abnormal Liver Functions: Bilirubin more 3 mg/dL, transaminases (AST/ALT) more than 2.5 times the institutional upper limits of normal (IULN).
* Systemic active infection, unless controlled on active therapy.
* Patients with Grade III/IV cardiac problems as defined by the New York Heart Association (NYHA) Criteria ( i.e., congestive heart failure, myocardial infarction within 6 months of the study), or ejection fraction (EF)< 30%.
* Patient has known chronic liver disease (i.e., chronic active hepatitis, hepatitis B, hepatitis C, and cirrhosis).
* Patient has known diagnosis of human immunodeficiency virus (HIV) infection.
* History of other malignancy, except non-melanotic skin cancers or no disease recurrence/progression for more than 2 years.
* Patients that have received investigational agents within 1 month of study entry.
* History of allergic reaction attributed to compounds of similar chemical or biologic composition to Gleevec or any component of the CLAG regimen
* Prior therapy with CLAG chemotherapy regimen
* Any adverse event attributable to previous chemotherapy regimen must be resolved to grade 1 or less at time of registration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2009-08; Primary Completion 2012-12 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rami Komrokji, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between August 2009 and April 2011, participants were enrolled at Moffitt Cancer Center.
Period: Overall Study
Arm/Group | CLAG Regimen With Gleevec®
Started | 38
Completed | 38
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | CLAG Regimen With Gleevec®
Number analyzed (Participants) | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 15
Age, Continuous [Median (Full Range); unit: years] | 62 [26 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 22
Region of Enrollment [Number; unit: participants]
  United States | 38

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: Overall Response Rate: Morphologic Complete Remission (CR) + Morphologic Complete Remission with incomplete blood count recovery (CRi) for evaluable participants. CR - Bone Marrow: < 5% blasts without Auer rods with at least 20% cellularity with maturation of all cell lines, No presence of unique phenotype by flow cytometry identical to what was found in the pretreatment specimen, No persistent dysplasia; Peripheral: normal blood counts, absolute neutrophil count (ANC) > 1.0 k/μl and platelets > 100 k/μl ANC > 1.0 k/μl and platelets > 100 k/μl (Peripheral blood counts documenting recovery can be utilized within 4 weeks of the bone marrow); No evidence of extramedullary leukemia. CRi - All CR criteria are met except for residual Neutropenia <1.0 x 10^9/L platelets < 100 k/μl.
Time Frame: 8 weeks per participant
Population: All participants
Measure: Number; unit: percentage of participants
Arm/Group | CLAG Regimen With Gleevec®
Number analyzed (Participants) | 38
percentage of participants | 37

2. Secondary Outcome: Median Progression Free Survival (PFS)
Description: Progression Free Survival is defined as the duration of time from start of treatment to time of progression. Leukemia related failure (progressive disease): Failure to induce bone marrow hypoplasia after 2 cycles or regrowth of leukemic blasts ≥ 20%.
Time Frame: Up to 3 years
Population: All participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | CLAG Regimen With Gleevec®
Number analyzed (Participants) | 38
months | 11.1 [4.8 to 13.4]

3. Secondary Outcome: Median Overall Survival (OS)
Description: Overall Survival is defined as the time from randomization until death from any cause.
Time Frame: Up to 3 years
Population: All participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | CLAG Regimen With Gleevec®
Number analyzed (Participants) | 38
months | 4.9 [1.6 to 11.7]

ADVERSE EVENTS:
Time Frame: 1 year, 10 months
Arm/Group | CLAG Regimen With Gleevec®
Serious Adverse Events (participants affected / at risk) | 8/38
Other Adverse Events (participants affected / at risk) | 38/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CLAG Regimen With Gleevec® (N=38)
Death not associated with CTCAE term - Disease progression NOS (General disorders) | 1 (1)
Hemorrhage, pulmonary/upper respiratory - Lung (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Liver dysfunction/failure (clinical) (Hepatobiliary disorders) | 1 (1)
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils - Blood (Infections and infestations) | 1 (1)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 1 (1)
Pain - Abdomen NOS (General disorders) | 1 (1)
Pain - Cardiac/heart (General disorders) | 1 (1)
Adult Respiratory Distress Syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thrombosis/embolism (vascular access-related) (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CLAG Regimen With Gleevec® (N=38)
Diarrhea (Gastrointestinal disorders) | 29 (30)
Nausea (Gastrointestinal disorders) | 28 (29)
Vomiting (Gastrointestinal disorders) | 20 (22)
Anorexia (Gastrointestinal disorders) | 12 (12)
Constipation (Gastrointestinal disorders) | 9 (10)
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 8 (8)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 3 (3)
Dehydration (Gastrointestinal disorders) | 2 (2)
Gastrointestinal - Other (Gastrointestinal disorders) | 2 (2)
Febrile neutropenia (Infections and infestations) | 22 (31)
Infection with Grade 3 or 4 neutrophils - Lung (pneumonia) (Respiratory, thoracic and mediastinal disorders) | 16 (18)
Infection with Grade 3 or 4 neutrophils - Blood (Infections and infestations) | 12 (12)
Infection - Other (Infections and infestations) | 10 (11)
Infection with Grade 3 or 4 neutrophils - Small bowel NOS (Infections and infestations) | 6 (6)
Infection with Grade 3 or 4 neutrophils - Urinary tract NOS (Infections and infestations) | 5 (5)
Infection with Grade 3 or 4 neutrophils - Colon (Infections and infestations) | 4 (4)
Infection with normal ANC or Grade 1 or 2 neutrophils - Lung (pneumonia) (Infections and infestations) | 3 (3)
Infection with normal ANC or Grade 1 or 2 neutrophils - Blood (Infections and infestations) | 2 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils - Mucosa (Infections and infestations) | 2 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils - Urinary tract NOS (Infections and infestations) | 2 (2)
Infection with Grade 3 or 4 neutrophils - Skin (cellulitis (Skin and subcutaneous tissue disorders) | 3 (3)
Infection with unknown AND - Lung (pneumonia) (Infections and infestations) | 2 (2)
Edema: limb (Blood and lymphatic system disorders) | 32 (35)
Lymphatics - Other (Blood and lymphatic system disorders) | 8 (8)
Edema: head and neck (Blood and lymphatic system disorders) | 2 (2)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 15 (17)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 11 (11)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 8 (8)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 8 (8)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 6 (6)
AST, SGOT (serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 5 (5)
Acidosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 3 (3)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 2 (2)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 2 (2)
Rigors/chills (General disorders) | 17 (24)
Insomnia (General disorders) | 7 (7)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 5 (5)
Constitutional Symptoms - Other (General disorders) | 2 (2)
Fever (in the absence of neutropenia) (General disorders) | 2 (2)
Sweating (diaphoresis) (General disorders) | 2 (2)
Weight gain (General disorders) | 2 (2)
Pain - Head/headache (General disorders) | 8 (8)
Pain - Back (General disorders) | 5 (5)
Pain - Abdomen NOS (General disorders) | 4 (4)
Pain - Extremity-limb (General disorders) | 4 (4)
Pain - Joint (General disorders) | 4 (5)
Pain-Cardiac/heart (General disorders) | 3 (3)
Pain - Chest/thorax NOS (General disorders) | 2 (2)
Pain - Neck (General disorders) | 2 (2)
Mood alteration - Anxiety (Psychiatric disorders) | 12 (12)
Confusion (Psychiatric disorders) | 7 (7)
Psychosis (hallucinations/delusions) (Psychiatric disorders) | 5 (6)
Mood alteration - Depression (Psychiatric disorders) | 4 (4)
Dizziness (General disorders) | 3 (3)
Memory impairment (General disorders) | 3 (3)
Mental status (Psychiatric disorders) | 3 (3)
Syncope (fainting) (General disorders) | 2 (2)
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 14 (14)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 6 (6)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 4 (4)
Rash: dermatitis associated with radiation - Chemoradiation (Skin and subcutaneous tissue disorders) | 3 (3)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 2 (2)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Adult Respiratory Distress Syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hemorrhage, pulmonary/upper respiratory - Nose (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Hemorrhage/Bleeding - Other (General disorders) | 4 (4)
Hemorrhage, GI - Lower GI NOS (Gastrointestinal disorders) | 3 (3)
Cardiac General - Other (Cardiac disorders) | 4 (5)
Hypertension (Cardiac disorders) | 3 (3)
Hypotension (Cardiac disorders) | 3 (3)
Cardiac troponin T (cTnT) (Cardiac disorders) | 2 (2)
Left ventricular systolic dysfunction (Cardiac disorders) | 2 (2)
Renal failure (Renal and urinary disorders) | 6 (6)
Renal/Genitourinary - Other (Renal and urinary disorders) | 2 (2)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 5 (5)
Dry eye syndrome (Eye disorders) | 3 (3)
Vision-blurred vision (Eye disorders) | 3 (3)
Ocular/Visual - Other (Eye disorders) | 2 (2)
Muscle weakness, generalized or specific area (not due to neuropathy) - Extraocular (Eye disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes